CLINICAL TRIAL: NCT04690712
Title: The Effect of Health Education Provided to Primary School Students on Screening Results
Brief Title: Health Education Provided to Primary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: KaratayBB
Record Dates: First submitted 2020-12-08; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Nurse's Role; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Health screening was done to the experimental group with one group. Surveys were conducted. Later, health education was given to this group. Six months later, the same group was screened for health again and a questionnaire was applied.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Socio-Demographic Characteristics of Students (No Intervention): When the socio-demographic characteristics of the students are examined according to the pre-test findings; It was seen that 27% were in the first grade, 20.9% in the second grade, and 25.7% in the third grade. When the age groups were evaluated, it was determined that 47.8% were in the 7-8 age group, 51.5% were in the 9-10 age group and 50% of them were female students and 50% were male students. It was observed that 27.6% of the students had a bad income and 59.3% had a medium level of income. When the father's education status was questioned, it was determined that 17.6% of them did not finish primary school, 55.4% of them were primary school graduates, 2.6% of them were high school graduates. On the other hand, 55% of their mothers did not complete primary school, 43.5% were primary school graduates and 1.5% were secondary school graduates
- Comparison of Students' Pretest and Posttest Development Screening Average (Experimental): According to the results of height and weight screening at the pre-test stage; the average height of the students is 127.0 ± 9.11; It was determined that the average weight was 26.1 ± 6.19, the average height was 130.61 ± 8.83 and the average weight was 29.92 ± 6.39 in the final test stage. A significant difference was found between pre-test and post-test screening results
  Interventions: Behavioral: Health Education
- Comparison of Pre-Test and Post-Test Screening Results of Students (Experimental): In the statistical evaluation, it was found that there was no significant difference between pre-test and post-test screening results
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — All students who attended the school were provided training by the researchers to improve oral and dental health and general hygiene. These trainings were made using slide shows and various entertaining materials. In addition, education was transformed into a drama with a theater show, and the importance of hand washing, hair and toilet hygiene was explained.
  In addition to hygiene, students were given training on correct eating patterns for a day so that they could develop healthy.
  Arms: Comparison of Pre-Test and Post-Test Screening Results of Students; Comparison of Students' Pretest and Posttest Development Screening Average

SUMMARY:
This study was conducted in a primary school in turkey.It was aimed to examine the effects of health education given to children in primary school period.As a result, it has been seen that education can be effective.

DETAILED DESCRIPTION:
Investigation of the Effects of Health Education Provided to Saraçoğlu Toki Mustafa Çetin Primary School Students on Health Screening Results The aim of this study is to find the effect of health education given to primary school students on health screening results.

The research is a pre-test and post-test quasi-experimental model with a single subject group. Saracoglu Toki Mustafa Cetin Primary School is that located in Turkey; It was held between September 2019 and March 2020. It was aimed to reach the entire universe, not choosing the sample. The pre-test screening was completed with 460 students and the post-test screening with 400 students. An Introductory Information Form and Screening Test Application Form were used to collect data. After the health education was given by the researchers using visual, auditory materials and drama technique, the results were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All students who regularly attend school at Saraçoğlu TOKI Primary School and who had no communication problems and whose parents gave their research approval were included in the study.

Exclusion Criteria:

* Students who could not attend school were excluded from the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Screening Tests Application Form | 6 months
  This form developed by the researchers by scanning the literature; It consists of a total of six screening phases including height, weight, oral hygiene, scalp hygiene / lice-dandruff and snellen / vision tests. It was used by the researchers to determine the results of the scan by selecting "yes", "no" options.
Introductory Information Form | 1 week
  While collecting the data, an Introductory Information Form developed by the researchers, consisting of eight questions including questions such as class, age, gender, family income, father's education level, mother's education status, father's occupation and mother's occupation, was used.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Dr Bayır, 1, Principal Investigator — KTO Karatay University
Locations (1):
- Berna Bayır, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No